CLINICAL TRIAL: NCT05047172
Title: Comparison of Anti-coagulation and Anti-Platelet Therapies for Intracranial Vascular Atherostenosis (CAPTIVA)
Brief Title: Comparison of Anti-coagulation and Anti-Platelet Therapies for Intracranial Vascular Atherostenosis
Acronym: CAPTIVA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Cincinnati (Other); Medical University of South Carolina (Other); Janssen Scientific Affairs, LLC (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CED000000522; AWD10099 (Other: UFIRST); U01NS117450 (NIH)
Record Dates: First submitted 2021-09-07; First posted 2021-09-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Arteriosclerosis; Stroke
MeSH Terms: conditions — Intracranial Arteriosclerosis; Stroke | interventions — Ticagrelor; Aspirin; Rivaroxaban; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 1:1:1 treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Experimental Arm: Ticagrelor and Aspirin (Experimental): Ticagrelor (180mg loading dose, then 90mg twice daily) and aspirin (81mg daily)
  Interventions: Drug: Ticagrelor + Aspirin; Other: Risk Factor Management
- Standard of Care Arm: Clopidogrel and Aspirin (Active Comparator): Clopidogrel (600mg loading dose, then 75mg once daily) and aspirin (81mg daily)
  Interventions: Drug: Clopidogrel + Aspirin; Other: Risk Factor Management
- Experimental Arm: Rivaroxaban and Aspirin (Experimental): Rivaroxaban (2.5mg twice daily) and aspirin (81mg daily)
  Interventions: Drug: Rivaroxaban + Aspirin; Other: Risk Factor Management

INTERVENTIONS:
Drug: Ticagrelor + Aspirin — ticagrelor (180 mg loading dose, then 90mg twice daily) and aspirin (81mg daily)
  Other Names: Brilinta
  Arms: Experimental Arm: Ticagrelor and Aspirin
Drug: Rivaroxaban + Aspirin — low dose rivaroxaban (2.5mg twice daily) and aspirin (81mg daily)
  Other Names: Xarelto
  Arms: Experimental Arm: Rivaroxaban and Aspirin
Drug: Clopidogrel + Aspirin — clopidogrel (600mg loading dose, then 75mg daily) and aspirin (81mg daily)
  Other Names: Plavix
  Arms: Standard of Care Arm: Clopidogrel and Aspirin
Other: Risk Factor Management — Risk factors for stroke (LDL, blood pressure, non-HDL cholesterol, diabetes, smoking, weight, and physical activity) will be monitored and managed.

SUMMARY:
The primary goal of the trial is to determine if the experimental arms (rivaroxaban or ticagrelor or both) are superior to the clopidogrel arm for lowering the 1-year rate of ischemic stroke, intracerebral hemorrhage, or vascular death.

DETAILED DESCRIPTION:
The proposed study is relevant to public health because narrowing of brain arteries is one of the most common causes of stroke worldwide. Compelling evidence suggests novel antithrombotic medications could reduce the rate of stroke in patients with narrowed brain arteries. The proposed study will directly compare novel antithrombotic medications to standard care antiplatelet medications for preventing stroke and death from vascular causes in patients with narrowed brain arteries.

ELIGIBILITY:
Inclusion Criteria:

* Acute focal symptoms or signs of any duration associated with imaging, pathological, or other objective evidence of arterial infarction OR clinical evidence of cerebral, spinal cord, or retinal focal arterial ischemic injury based on symptoms persisting greater than or equal to 24 hours that occurred within 30 days prior to randomization
* Index stroke is attributed to 70-99% stenosis (or flow gap on MRA) of a major intracranial artery (carotid artery, middle cerebral artery (M1 or M2), vertebral artery (V4), basilar artery, posterior cerebral artery (P1), or anterior cerebral artery (A1)) documented by CTA, MRA, or catheter angiography
* Modified Rankin Scale score of ≤ 4, at time of consent
* Ability to swallow pills
* At least 30 years of age, inclusive, at time of consent
* Subjects 30-49 years of age are required to meet at least ONE of the following additional criteria below to qualify for the study:

  1. diabetes treated with insulin for at least 15 years
  2. at least 2 of the following atherosclerotic risk factors: hypertension (BP > 140/90 or on antihypertensive therapy); dyslipidemia (LDL > 130 mg /dl or HDL < 40 mg/dl or fasting triglycerides > 150 mg/dl or on lipid lowering therapy); smoking; non-insulin dependent diabetes or insulin dependent diabetes of less than 15 years duration; any of the following vascular events occurring in a parent or sibling who was < 55 years of age for men or < 65 years of age for women at the time of the event: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, stroke, carotid endarterectomy or stenting, peripheral vascular surgery for atherosclerotic disease
  3. personal history of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, carotid endarterectomy or stenting, or peripheral vascular surgery for atherosclerotic disease
  4. any stenosis of an extracranial carotid or vertebral artery, another intracranial artery, subclavian artery, coronary artery, iliac or femoral artery, other lower or upper extremity artery, mesenteric artery, or renal artery that was documented by non-invasive vascular imaging or catheter angiography and is considered atherosclerotic
  5. aortic arch atheroma documented by non-invasive vascular imaging or catheter angiography
  6. any aortic aneurysm documented by non-invasive vascular imaging or catheter angiography that is considered atherosclerotic
* Negative pregnancy test in a female who has had any menses in the last 18 months and has not had surgery that would make her unable to become pregnant
* Subject is willing and able to return for all follow-up evaluations required by the protocol
* Subject is available by phone
* Subject understands the purpose and requirements of the study and can make him/herself understood
* Subject has provided informed consent (use of a LAR is not permitted)

Exclusion Criteria:

* Previous treatment of qualifying intracranial artery with a stent, angioplasty, or other mechanical device, including mechanical thrombectomy for the qualifying stroke, or plan to perform one of these procedures
* Plan to perform concomitant endarterectomy, angioplasty or stenting of an extracranial vessel tandem to the symptomatic intracranial stenosis
* Intracranial tumor (except meningioma) or any intracranial vascular malformation
* Thrombolytic therapy within 24 hours prior to randomization
* Progressive neurological signs within 24 hours prior to randomization
* History of spontaneous non-traumatic intracranial hemorrhage (parenchymal, subarachnoid, subdural, epidural)
* Intracranial arterial stenosis due to: arterial dissection; MoyaMoya disease; any known vasculitic disease; herpes zoster, varicella zoster or other viral vasculopathy; neurosyphilis; any other intracranial infection; any intracranial stenosis associated with CSF pleocytosis; radiation induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; benign angiopathy of central nervous system; postpartum angiopathy; suspected vasospastic process; reversible cerebral vasoconstriction syndrome (RCVS); suspected recanalized embolus
* Presence of any of the following unequivocal cardiac sources of embolism: chronic or paroxysmal atrial fibrillation, mitral stenosis, mechanical valve, endocarditis, intracardiac clot or vegetation, myocardial infarction within three months, left atrial spontaneous echo contrast
* Known allergy or contraindication to aspirin, rivaroxaban, clopidogrel, or ticagrelor
* Uncontrolled severe hypertension (systolic pressure > 180 mm Hg or diastolic pressure > 115 mm Hg), active peptic ulcer disease, major systemic hemorrhage within 30 days prior to randomization, active bleed or bleeding diathesis, platelets < 100,000, hematocrit < 30, INR > 1.5, clotting factor abnormality that increases the risk of bleeding, current alcohol or substance abuse, severe liver impairment (AST or ALT > 3 x normal, cirrhosis), or CrCl < 15 mL/min or on dialysis
* Major surgery (including stenting of any vessel; open femoral, aortic, or carotid surgery; or cardiac surgery) within previous 30 days prior to randomization or planned in the next 90 days after randomization
* Any condition other than intracranial arterial stenosis that requires the subject to take any antithrombotic medication other than aspirin (NOTE: exceptions allowed for subcutaneous heparin or enoxaparin for deep vein thrombosis (DVT) prophylaxis)
* Dementia or psychiatric problem that prevents the subject from following an outpatient program reliably
* Co-morbid conditions that may limit survival to less than 12 months
* Pregnancy or of childbearing potential and unwilling to use contraception for the duration of this study, or currently breastfeeding
* Current or anticipated concomitant oral or intravenous therapy with strong CYP3A4 inhibitors or CYP3A4 substrates that cannot be stopped for the course of this study
* Enrollment in another study that would conflict with the current study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1683 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with parenchymal ICH or non-ICH major hemorrhage | Up to 12 months
  Non-ICH major hemorrhage is derived from the International Society on Thrombosis and Haemostasis (ISTH) criteria consisting of any of the following:
  * Fatal bleeding
  * Symptomatic bleeding in a critical area or organ, such as subarachnoid, intraventricular, subdural, epidural, spinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome
  * Symptomatic bleeding causing a fall in hemoglobin level of 1.24 mmol/L (20g/L or greater) or more, or leading to transfusion of two units or more of whole blood or red cells
Number of participants with ischemic stroke, intracerebral hemorrhage or vascular death | Up to 12 months
  The definition of ischemic stroke is the American Heart Association definition that includes acute focal signs or symptoms of cerebral, spinal cord, or retinal involvement of any duration associated with imaging, pathological, or other objective evidence of arterial infarction OR clinical evidence of cerebral, spinal cord, or retinal focal arterial ischemic injury based on symptoms persisting greater than or equal to 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Brian L. Hoh, MD, MBA, Principal Investigator — University of Florida; Marc I. Chimowitz, MBChB, Principal Investigator — Medical University of South Carolina
Locations (117):
- United States (117):
  - University of Alabama Hospital, Birmingham, Alabama
  - University of South Alabama University Hospital, Mobile, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - Mercy San Juan Medical Center, Carmichael, California
  - The Neuron Clinic - Chula Vista, Chula Vista, California
  - Kaiser Permanente Fontana Medical Center, Fontana, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Los Alamitos Medical Center, Los Alamitos, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, CA, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - UC Davis Medical Center, Sacramento, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - UCSD Medical Center - Hillcrest Hospital, San Diego, California
  - Providence Little Company of Mary Medical Center Torrance, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - St. Mary's Medical Center, Grand Junction, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - UF Health Shands Hospital, Gainesville, Florida
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Cleveland Clinic Tradition Hospital, Port Saint Lucie, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Endeavor Health Edward Hospital, Naperville, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Javon Bea Hospital - Riverside, Rockford, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky Hospital, Lexington, Kentucky
  - Ochsner Medical Center - Main Campus, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Flint, Flint, Michigan
  - McLaren Macomb, Mount Clemens, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - M Health Fairview Southdale Hospital, Edina, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Health Care, Columbia, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Kings County Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - Buffalo General Medical Center, Buffalo, New York
  - North Shore University Hospital, Lake Success, New York
  - NYP Weill Cornell Medical Center, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - NYP Columbia University Medical Center, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - ECU Health Medical Center, Greenville, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Akron General, Akron, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - UH Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - OU Medical Center, Oklahoma City, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina University Hospital, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Covenant Medical Center, Lubbock, Texas
  - Medical City Plano, Plano, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - UT Health Tyler, Tyler, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - UVA Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Swedish Medical Center - Cherry Hill Campus, Seattle, Washington
  - University of Wisconsin University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No